CLINICAL TRIAL: NCT04000503
Title: Integrated Cervical Cancer Screening in Mayuge District Uganda (ASPIRE Mayuge): A Pragmatic Cluster Randomized Control Trial
Brief Title: Integrated Cervical Cancer Screening in Mayuge District Uganda (ASPIRE Mayuge)
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Uganda Cancer Institute (Other)
Responsible Party: Principal Investigator, Gina Ogilvie, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H17-03332
Record Dates: First submitted 2019-06-18; First posted 2019-06-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Human Papillomavirus 16; Human Papillomavirus 18; Papillomavirus Infections; Cervical Cancer; Pre-Cancerous Dysplasia
Keywords: Human Papillomavirus DNA Tests; Visual inspection with acetic acid; Global Health; Developing Countries; Self-collection; Cervical Cancer Screening
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Pragmatic cluster randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker Self-Collection (Experimental): Door-to-door recruitment of women for self-collected HPV testing
  Interventions: Behavioral: Self-collected HPV testing for cervical cancer screening
- Community Health Meeting Self-Collection (Experimental): Community health meeting recruitment of women for self-collected HPV testing
  Interventions: Behavioral: Self-collected HPV testing for cervical cancer screening

INTERVENTIONS:
Behavioral: Self-collected HPV testing for cervical cancer screening — Self-collection cervical cancer screening, STI screening, and education on HIV by a community health worker. Women who test positive for high-risk HPV types will be referred to a designated health centre for VIA follow-up and treatment if indicated.

SUMMARY:
The purpose of this pragmatic cluster randomized control trial is to test the effectiveness of cervical cancer screening follow-up completion using two implementation approaches for self-collected HPV testing in a rural, low-resource setting: 1) community health workers recruiting women door-to-door and 2) community health workers recruiting women at community health meetings.

This study will also help to further understand how current patient referral systems are working between health facilities, patient and provider preferences for integrated care and health system related barriers to integrated cervical cancer screening.

Hypothesis: More women will receive screening via the community health meeting but the engagement to care (i.e., visual inspection with acetic acid-our main outcome) will be greater in the door-to-door arm.

DETAILED DESCRIPTION:
A cluster randomized control trial will be conducted with the objective of understanding differences in the effectiveness of cervical cancer screening models using self-collected HPV testing on engagement in care. In 31 villages, women will be recruited for self-collected cervical cancer and sexually transmitted infection (STI) screening by: 1) Community health worker recruitment for self-collection (door-to-door), 2) community health meetings. Visual inspection with acetic acid (VIA), cryotherapy and thermocoagulation will be offered in local health facilities for all women who test positive for high-risk (HR)-HPV types. Women needing advanced cancer care will be referred to the Uganda Cancer Institute in Kampala.

The unit of randomization (2 arms) will be villages and the analysis will also account for clustering within this unit or randomization. All participants will receive an integrated package of cervical cancer screening and education and will participate in a survey at baseline. Samples will be tested using GeneXpert (XpertHPV) point of care testing at the Kigandalo health facility for HPV and high risk HPV (HR-HPV). Intervention arms will be implemented in phases by year to avoid temporal contamination.

ELIGIBILITY:
Inclusion Criteria:

* Women with no previous history of hysterectomy
* aged 25-49 years old
* no previous history of treatment for cervical cancer
* provided written informed consent.

Exclusion Criteria:

* Women who are under 25 or over 49 years of age,
* who have previously had a hysterectomy or been treated for cervical cancer
* unable to provided informed consent.

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2019 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
VIA follow-up and treatment when indicated (screen and treat) | Outcome measured within 6 weeks of self-collection for HPV test
  Proportion of total screened women who complete VIA follow-up and treatment after testing positive for high-risk HPV type

SECONDARY OUTCOMES:
HPV prevalence | Baseline
  Total number of women who test positive for HPV out of the total number of samples obtained
STI-HPV co-infection rate (Gonorrhea, Syphilis, etc.) | Baseline
  Total number of women who test positive for STIs out of total number of women who test positive for HPV; total number of women who test negative for STIs out of total number of women who test positive for HPV; total number of women who test positive for STIs out of total number of women who test negative for HPV; total number of women who test negative for STIs out of total number of women who test negative for HPV
HPV and co-morbid conditions | Baseline
  Association (adjusted OR) estimated between HPV and HIV; other STIs
Barriers and facilitators of engagement in care | FGDs within 3 months of recruitment completion
  Semi-structured focus group discussions with women who did and did not attend follow-up screening in each study arm.
Identify mediators of engagement of care | Outcome measured within 6 weeks of self-collection for HPV test
  Mediation analysis using counterfactual approach to assess mediating effect of patient reported experience, knowledge change and co-infection status with other STIs on engagement in care after positive HR-HPV test

OTHER OUTCOMES:
Cost-effectiveness of each model of community-based cervical cancer screening | Modeled lifetime estimates after 1 year follow-up
  Measured using years of lives saved compared between each study arm and the ICER
Process evaluation for integrated community-based cervical cancer screening | Within 6 months of final recruitment
  Evaluating reach, fidelity, barriers and facilitators of implementation in each arm from the community and health system perspective using mixed methods
Male partner knowledge of cervical cancer screening | Baseline
  Assess men's knowledge level of HPV and cervical cancer and determine which factors impact the supportiveness towards a partner seeking screening.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Ogilvie, MD, Principal Investigator — Women's Health Research Institute of British Columbia; Sheona Mitchell-Foster, MD, Principal Investigator — University of Northern British Columbia; Carolyn Nakisige, MD, Principal Investigator — Uganda Cancer Institute
Locations (1):
- Uganda Cancer Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
Data will be available on request through study investigators.

REFERENCES:
- [Derived] Leahy W, Abomoslim M, Booth A, Gottschlich A, Mwandacha N, Dau H, Naguti P, Payne B, Smith L, Nakisige C, Ogilvie G. Women's cellphone access and ownership in rural Uganda: implications for self-care interventions. BMC Glob Public Health. 2024 Feb 5;2(1):8. doi: 10.1186/s44263-024-00038-5. PMID 39681893
- [Derived] Gottschlich A, Payne BA, Trawin J, Albert A, Jeronimo J, Mitchell-Foster S, Mithani N, Namugosa R, Naguti P, Pedersen H, Rawat A, Simelela PN, Singer J, Smith LW, van Niekerk D, Orem J, Nakisige C, Ogilvie G. Community-integrated self-collected HPV-based cervix screening in a low-resource rural setting: a pragmatic, cluster-randomized trial. Nat Med. 2023 Apr;29(4):927-935. doi: 10.1038/s41591-023-02288-6. Epub 2023 Apr 10. PMID 37037880
- [Derived] Gottschlich A, Payne BA, Trawin J, Albert A, Jeronimo J, Mitchell-Foster S, Mithani N, Namugosa R, Naguti P, Orem J, Rawat A, Simelela PN, Singer J, Smith LW, van Niekerk D, Nakisige C, Ogilvie G. Experiences with thermal ablation for cervical precancer treatment after self-collection HPV-based screening in the ASPIRE Mayuge randomized trial. Int J Cancer. 2023 Apr 15;152(8):1630-1639. doi: 10.1002/ijc.34369. Epub 2022 Nov 28. PMID 36408923
- [Derived] Rawat A, Mithani N, Sanders C, Namugosa R, Payne B, Mitchell-Foster S, Orem J, Ogilvie G, Nakisige C. "We Shall Tell them with Love, Inform them what we have Learnt and then Allow them to go" - Men's Perspectives of Self-Collected Cervical Cancer Screening in Rural Uganda: A Qualitative Inquiry. J Cancer Educ. 2023 Apr;38(2):618-624. doi: 10.1007/s13187-022-02163-x. Epub 2022 Apr 6. PMID 35384556
- [Derived] Nakisige C, Trawin J, Mitchell-Foster S, Payne BA, Rawat A, Mithani N, Amuge C, Pedersen H, Orem J, Smith L, Ogilvie G. Integrated cervical cancer screening in Mayuge District Uganda (ASPIRE Mayuge): a pragmatic sequential cluster randomized trial protocol. BMC Public Health. 2020 Jan 31;20(1):142. doi: 10.1186/s12889-020-8216-9. PMID 32005202